CLINICAL TRIAL: NCT06856564
Title: Evaluation of Tongue Mobility in Patients with Ankyloglossia Following Frenectomy
Brief Title: Tongue Mobility in Patients with Ankyloglossia Following Frenectomy
Status: Completed | Type: Observational
Sponsor: Hanoi Medical University (Other)
Responsible Party: Principal Investigator, Nguyen Ngoc Hoa, DDS, MDS, Hanoi Medical University
Other Study IDs: 1104
Record Dates: First submitted 2025-02-19; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Ankyloglossia
MeSH Terms: conditions — Ankyloglossia | interventions — Oral Frenectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Frenectomy — The study involves using a diode laser and scalpel to treat ankyloglossia in cases that are unresponsive to tongue exercises or exhibit severe restrictions. The techniques employed range from simple frenotomy to complex frenuloplasty, depending on the severity of the condition. Electrocautery is frequently used to minimize bleeding, although it may result in scar formation.

SUMMARY:
This study aimed to evaluate the improvement in tongue mobility in patients with ankyloglossia (tongue-tie) following frenectomy. Ankyloglossia restricts tongue movement, potentially causing issues with speech, swallowing, and dental malocclusion.

ELIGIBILITY:
Inclusion Criteria:

* (1) at least four years of age, (2) report a limitation in tongue mobility at least at the moderate class (class II) according to Kotlow criteria and did not response to tongue lengthening exercise.

Exclusion Criteria:

* Patients who have limited mouth openings that interfere with tongue mobility measurements and patients who have bad compliances due to mental problems or uncooperative children were excluded.

Ages: 4 Years to 33 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients at Hanoi National Hospital of Odonto-stomatology and Hanoi Medical University from December 2022 to December 2024
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Kotlow index | 3 months
  The Kotlow index measures the distance point of attachment of the frenum on the ventral surface of the tongue and the tip of the tongue. This outcome measure will be assessed in millimeters (mm) using the Quick Tongue-Tie (QTT) Assessment Tool.
Tongue-Incisive Papilla Distance | 3 months
  Tongue-Incisive Papilla (TIP) Distance is the distance between Tongue and Incisive Papilla. Ask the patient to open their mouth and simultaneously keep tongue tip touching the upper central papilla, the distance between upper and lower right central incisors is defined as TIP. This outcome measure will be assessed in millimeters (mm) using the Quick Tongue-Tie (QTT) Assessment Tool.
Comfortable Mouth Opening | 3 months
  Comfortable Mouth Opening (CMO) is the optimal jaw position during relaxed oral function, measured as the distance between the upper and lower teeth when the patient siting in upright posture, being relax and looking straight forward, and the mouth is naturally open. This outcome measure will be assessed in millimeters (mm) using the Quick Tongue-Tie (QTT) Assessment Tool.
Lingual - Palatal Suction | 3 months
  Lingual - Palatal Suction (LPS) is the distance between the upper and lower right central incisors when opening while the tongue is elevated to touch the hard palate. This outcome measure will be assessed in millimeters (mm) using the Quick Tongue-Tie (QTT) Assessment Tool.

CONTACTS AND LOCATIONS:
Locations (1):
- Hanoi National Hospital of Odonto-Stomatology, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes